CLINICAL TRIAL: NCT02152137
Title: A Phase 2 Study of Efatutazone, an Oral PPAR Agonist, In Combination With Paclitaxel in Patients With Advanced Anaplastic Thyroid Cancer
Brief Title: Inolitazone Dihydrochloride and Paclitaxel in Treating Patients With Advanced Anaplastic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A091305; U10CA031946 (NIH); U10CA180821 (NIH); NCI-2014-00686 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anaplastic Thyroid Cancer; Recurrent Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — efatutazone; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- efatutazone dihydrochloride, paclitaxel (Experimental): Patients receive paclitaxel IV over 3 hours on day 1 and efatutazone dihydrochloride PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: efatutazone; Drug: paclitaxel

INTERVENTIONS:
Drug: efatutazone — Given PO
  Other Names: CS-7017
Drug: paclitaxel — Given IV
  Other Names: Taxol

SUMMARY:
This phase II trial studies how well inolitazone dihydrochloride (efatutazone dihydrochloride) and paclitaxel work in treating patients with anaplastic thyroid cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Drugs used in chemotherapy, such as efatutazone dihydrochloride and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the combination of paclitaxel and efatutazone (efatutazone dihydrochloride) improves the confirmed response rate in patients with advanced anaplastic thyroid cancer.

SECONDARY OBJECTIVES:

I. To estimate the overall survival (OS), duration of response, progression-free survival (PFS), and adverse event rates for the combination of paclitaxel and efatutazone.

TERTIARY OBJECTIVES:

I. The association of biomarkers with clinical outcome data will be assessed in an exploratory translational analysis.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 3 hours on day 1 and efatutazone dihydrochloride orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 28 days, every 8 weeks until disease progression, and then every 6 months for 5 years.

ELIGIBILITY:
* Patients must have histologically or cytologically diagnosed advanced anaplastic thyroid cancer (ATC)
* Patients must have measurable disease
* Patients must have either metastatic (stage IVC) or locally advanced unresectable disease (stage IVB)
* Patients should have resolution of any toxic effects of prior therapy (except alopecia) to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, grade 1
* There is no limit to the number of prior lines of treatment a patient has received
* No treatment with chemotherapy, radiation therapy, immunotherapy, biological therapy, hormonal therapy, or other thiazolidinediones (TZDs) =< 21 days before study registration
* No prior taxane therapy =< 6 months, except as a radiosensitizer
* No history of the following:

  * Class III or IV congestive heart failure (CHF)
  * Grade 3 or 4 thromboembolic event =< 6 months
  * Pericardial effusion =< 12 months (any grade)
  * Pericardial involvement with tumor
  * Grade 2 or higher pleural effusion =< 6 months
* No current symptomatic, untreated, or uncontrolled brain metastases present
* No major surgery =< 14 days prior to registration
* No grade 2 or higher neuropathy
* No known history of severe hypersensitivity reactions to any of the components of efatutazone or paclitaxel formulations
* Not pregnant and not nursing; women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Patients with diabetes mellitus requiring concurrent treatment with insulin or thiazolidinedione (TZD) oral agents are not eligible
* Patients with known hypersensitivity to any TZD oral agents are not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN) mg/dL OR calculated (calc.) creatinine clearance >= 60 mL/min
* Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Although they will not be considered formal eligibility (exclusion) criteria, physicians should recognize that the following may seriously increase the risk to the patient entering this protocol:

  * Psychiatric illness which would prevent the patient from giving informed consent
  * Medical condition such as uncontrolled infection (including human immunodeficiency virus [HIV]), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
  * Patients with a "currently active" second malignancy other than non-melanoma skin cancers; patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years; there is an exception for patients with a history of well differentiated thyroid cancer that has progressed to anaplastic thyroid cancer
  * Patients who cannot swallow oral formulations of the agent(s)
  * Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study ; appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom)
  * Efatutazone is metabolized by cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5), and inhibits CYP2C8, 2C9, 2C19, and 3A4, and is a substrate of P-glycoprotein (PgP) and breast cancer resistance protein (BCRP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smallridge, M.D., Study Chair — Mayo Clinic
Locations (253):
- United States (253):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University Pointe, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Cabanillas ME, McFadden DG, Durante C. Thyroid cancer. Lancet. 2016 Dec 3;388(10061):2783-2795. doi: 10.1016/S0140-6736(16)30172-6. Epub 2016 May 27. PMID 27240885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients assigned to arm A will receive both paclitaxel and efatutazone; patients assigned to arm B will receive paclitaxel alone. However, please note that with update #2, arm B is closed and all patients should receive paclitaxel and efatutazone.
Groups:
- Efatutazone Dihydrochloride, Paclitaxel: Patients receive 175 mg/m^2 paclitaxel IV over 3 hours on day 1 and 0.5 mg efatutazone dihydrochloride PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Started (Enrolled) | 19
Originally Assigned to Arm A | 16
Originally Assigned to Arm B | 3 (With update #2, Arm B is closed and all patients should receive paclitaxel and efatutazone.)
Completed (received efatutazone and paclitaxel combination and were included in safety and efficacy analyses) | 15
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Originally assigned to Arm B | 3

BASELINE CHARACTERISTICS:
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 4
    1 | 9
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Partial Response [PR] or Complete Response [CR]) Per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 Criteria
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: Up to 24 weeks
Population: Patients who received efatutazone and paclitaxel combination were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 15
percentage of patients | 13 [2 to 40]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from study entry to death from any cause, assessed up to 5 years
Population: Patients who received efatutazone and paclitaxel combination were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 15
months | 6.6 [4.2 to 27.3]

3. Secondary Outcome: Duration of Confirmed Response
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression (PD) is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir).
Time Frame: The time from the first documented date of confirmed response (CR or PR) to date at which progression is first documented, assessed up to 5 years
Population: Only patients who achieved a confirmed response are included in this analysis.
Measure: Number; unit: months
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 2
months
  Patient #1 | 12.2
  Patient #2 | 3.2

4. Secondary Outcome: PFS Determined Based on RECIST 1.1 Criteria
Description: Progression free survival (PFS) is defined as the time from the date of registration to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The time from study entry to the first of either disease progression or death from any cause, assessed up to 5 years
Population: Patients who received efatutazone and paclitaxel combination were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 15
months | 2.5 [1.2 to 6.3]

5. Secondary Outcome: Number of Patients Experiencing at Least One Grade 3+ Adverse Event Using CTCAE Version 4.0
Description: The number of patients who experienced at least one grade 3 or higher adverse event is reported below.
Time Frame: Up to 5 years
Population: Patients who received efatutazone and paclitaxel combination were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
Number analyzed (Participants) | 15
Participants | 13

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Evaluable patients who received efatutazone and paclitaxel combination and had adverse events assessed are summarized below.
Arm/Group | Efatutazone Dihydrochloride, Paclitaxel
All-Cause Mortality (participants affected / at risk) | 12/15
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efatutazone Dihydrochloride, Paclitaxel (N=15)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Neck edema (General disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efatutazone Dihydrochloride, Paclitaxel (N=15)
Anemia (Blood and lymphatic system disorders) | 12 (45)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (3)
Bloating (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (8)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (14)
Nausea (Gastrointestinal disorders) | 5 (21)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 1 (2)
Edema face (General disorders) | 2 (5)
Edema limbs (General disorders) | 10 (51)
Fatigue (General disorders) | 9 (29)
Fever (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Blood bilirubin increased (Investigations) | 2 (6)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (5)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (7)
Neutrophil count decreased (Investigations) | 6 (17)
Platelet count decreased (Investigations) | 3 (6)
Weight gain (Investigations) | 9 (36)
White blood cell decreased (Investigations) | 6 (21)
Anorexia (Metabolism and nutrition disorders) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (3)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (50)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (14)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (8)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (3)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT02152137/Prot_SAP_000.pdf